CLINICAL TRIAL: NCT00481117
Title: Safety, Tolerability, PK and PD of LY2405319 After Multiple Subcutaneous Injections in Subjects With Type 2 Diabetes
Brief Title: Safety, Tolerability, and Effect of LY2405319 After Multiple Injections in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 11719; I1K-MC-GLUD (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-05-31; First posted 2007-06-01 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2010-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LY2405319

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: LY2405319
Drug: Placebo

SUMMARY:
This study intends to evaluate how safe and well tolerated the LY2405319 compound is when given to people for 7 days (in Part 1) and 28 days (in Part 2). This study intends to also determine if there is a positive effect on lowering the level of glucose in people with type 2 diabetes.

DETAILED DESCRIPTION:
Subjects in Part 1 will be randomized to receive LY2405319 or placebo over 7 days in one of 4 dose level groups, in ascending order: 1 mg, 3 mg, 10 mg, or 20 mg.

Subjects in Part 2 will be randomized to receive LY2405319 or placebo over 28 days, and will receive the dose level determined to be the most well tolerated in Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Men and women without child bearing capability
* Ages 35 to 70 years
* Type 2 diabetic subjects, diagnosed for at least 3 months
* Average body weight (relative to height)
* Willing to be available for the duration of the study

Exclusion Criteria:

* Significant medical illnesses (except Type 2 diabetes)
* Abnormal 12-lead electrocardiogram (ECG )
* Current or previous use of insulin for greater than 7 days for control of diabetes
* Regular use of drugs of abuse
* Excessive alcohol use

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-08; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Safety labs, ECGs, vital signs, adverse events. | End of dosing period

SECONDARY OUTCOMES:
Pharmacodynamics (lab samples) and Pharmacokinetics (lab samples) | End of dosing period

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (11):
- India (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ambawadi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belagavi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabaad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maharashtra
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rabale
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Siddhapudur
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morelia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wellington, New Zealand
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., George, South Africa

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com